CLINICAL TRIAL: NCT06792617
Title: Exercise Rehabilitation in Patients With Severe Cardiopulmonary Dysfunction on Extracorporeal Life Support
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute for Extracorporeal Life Support (Other)
Responsible Party: Principal Investigator, Linda Sousse, Director of Research, Institute for Extracorporeal Life Support
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERECLS-01
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: ExtraCorporeal Membrane Oxygenation (ECMO); Cardiopulmonary Function; Rehabilitation
Keywords: Extracorporeal membrane oxygenation (ECMO); Rehabilitation exercise program
MeSH Terms: interventions — Range of Motion, Articular; Multicenter Studies as Topic; Resistance Training

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a prospective clinical trial on eligible adults (≥18 years) with severe cardiac and/or lung dysfunction placed on ECMO. Results will be compared to historical controls from MHS who have not been enrolled in a rehabilitation program, which is the current standard of care (SOC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Exercise Group (Other): The exercise group will complete the highest intensity exercise and activity as tolerated to maximize their progression of strength, function, and out of bed.
  This group will also be utlizing the VitalGo Total Lift Bed (TLB) V5 for vertical positioning to provide a better potential for hemodynamic response to activities to include: strength training, mobility tasks, and functional activities like Activities of Daily Living (ADL).
  Interventions: Other: Mobility (Central or Femoral Cannulation); Other: Resistance Training

INTERVENTIONS:
Other: Mobility (Central or Femoral Cannulation) — Functional Mobility & ADL's
  1. Assisted sitting with progression to unassisted; ADL's
  2. Assisted standing with progression to unassisted; ADL's
     1. VitalGo bed will be used if unsafe/unable to perform assisted standing.
     2. Leg press (VitalGo bed)
  3. Ambulation; ADL's
Other: Resistance Training — Repetitions will be counted and documented per session per structured exercise.

SUMMARY:
Short-term and long-term consequences of severe cardiac and/or lung dysfunction can be increased use of sedation, prolonged bedrest and immobility causing severe loss of muscle mass which could be a risk for muscle weakness, osteoporosis, and lowered endurance. The goal of this study is to show how a structured rehabilitation program can exhibit better short-term and long-term outcomes on patients who are treated with extracorporeal membrane oxygenation (ECMO).

DETAILED DESCRIPTION:
I.Introduction

The long-term consequences of severe cardiac and/or lung dysfunction include: the increased use of sedation, increased parameters on the ventilator, and incidence of delirium. These sequelae are all associated with prolonged bed rest and immobility, which causes severe loss of muscle mass and bone density. Significant loss of muscle and bone causes patients to be at risk for muscle weakness, osteoporosis, and lowered endurance. Extracorporeal membrane oxygenation (ECMO) is a strategy used to mitigate severe cardiac and/or lung dysfunction. Briefly, during ECMO, blood passes through a mechanical circuit and external oxygenator, which removes carbon dioxide and adds oxygen. Blood is then re-infused by a pump to provide cardiovascular support upon return to the body. It provides gas exchange for patients when their own heart and/or lungs are unable to function adequately, and it has been shown to improve survival rates and outcomes in patients with severe respiratory failure.

The investigators hypothesize that patients with cardiac and/or lung dysfunction treated with ECMO who participate in this rehabilitation program will exhibit better short-term and long-term outcomes than patients who have not participated in this rehabilitation program. There are four aims to this study: patients who participate in this rehabilitation program will exhibit a (1) significantly increased rate of weaning from ECMO and from mechanical ventilation, (2) significantly decreased rate of major post-ECMO complications, (3) significantly increased time exercising and improvement and completion of activities of daily living [ADL], and (4) significant increase in quality of life, long-term outcomes, short physical performance battery, and rehabilitation outcomes.

II. Background This study's intended accomplishment will be to establish a multidisciplinary, structured exercise and rehabilitation program for patients on ECMO so that days on an ECMO circuit are reduced, quality of life is improved, post-ECMO complications are decreased, and positive long-term outcomes are increased. This is important because there is no standard of care established for a structured exercise program for patients on ECMO. These patients are primarily bed bound for the majority of their illness in the early stages; if early implementation of a structured exercise regimen is started then the amount of time it takes patients to return to their physical physiological baseline will be decreased, thus improving their quality of life.

A thorough review of the literature indicates that there is a critical lack of studies of rehabilitation, movement, or physical activity in the ECMO patient population. Furthermore, a structured rehabilitation program for ECMO patients simply does not exist. The use of a structured resistant exercise program in this population has not been studied. Thus, overcoming this deficiency is extremely important for the 10% of intensive care unit (ICU) admissions with cardiac and respiratory failure across the nation, specifically those who are placed on ECMO.

Approximately 30 studies exist in the literature that describe rehabilitation in the ECMO patient population. Briefly, these studies in adults with severe lung dysfunction have shown that participation in rehabilitation programs incorporating mobility training and physical (PT) and occupational therapy (OT) significantly improve functional and physiological outcomes and decrease muscle wasting, sedation requirements, and length of stay. The patients that participate in rehabilitation also increase endurance and have full stabilization of the cardiopulmonary system and full recovery of neurological functions. Most importantly, it has been shown that patients with severe lung dysfunction who enter a rehabilitation program decrease mortality, and they are more likely to be discharged home.

III. Rationale There is a need for randomized controlled trials to study methods for rehabilitation in the ECMO population, and this proposal serves as the first step towards that goal. The investigators firmly believe that the activities proposed here will beneficially impact the ECMO patient population by improving physiological responses, physical function, and psychosocial well-being. In bed-ridden and immobile adults, exercise and movement are important in reducing risk factors such as obesity, insulin resistance, and general deconditioning. The evidence base for this program can be found in both the basic and clinical science literature of several patient populations: adult and pediatric burns, geriatric and frail, bed rest and antigravity (via National Aeronautics and Space Administration [NASA] studies), post-cardiac arrest, and traumatic brain injury (TBI). Hence, the investigators have formed a team of thought leaders from these areas to create a personalized rehabilitation program in the ECMO population.

This study will advance our knowledge in how a structured exercise program effects ECMO patients in their short- and long-term outcomes. There will be an advancement of knowledge in the physiological benefits of exercising ECMO patients. The verticalization into daily nursing care, mobility exercises, PT/OT, and resistance training will give the investigators a better understanding of the components that help keep muscle wasting minimal and help decrease a patient's length of stay.

Decreased muscle wasting and length of stay, decreased risk of mortality, and decreased sedation requirements will increase the likelihood that patients will have a full cardiopulmonary and neurological recovery. Longer treatment periods also translate into significant costs in dollars but, also in human cost/value.

SECTION B: RESEARCH PLAN

IV. Study Objectives The objectives of this study are to complete the highest intensity exercise and activity as tolerated by patients to maximize their progression of strength, function, and out of bed activity. In doing this, the investigators will also reduce the risk for potential of skin breakdown on common areas associated with decubitus pressure injuries and prolonged bedrest. In this study, the investigators will be utilizing the VitalGo Total Lift Bed (TLB) V5 for vertical positioning to provide a better potential for hemodynamic response to activities to include: strength training, mobility tasks, and functional activities like ADLs.

ELIGIBILITY:
Inclusion Criteria--

1. Age >or equal to 18 years old
2. On ECMO (VV and/or VA) for cardiopulmonary dysfunction/failure
3. Admitted to Lung Recovery Intensive Care Unit (LRICU) or Cardiovascular Intensive Care Unit (CVICU).
4. Richmond Agitation and Sedation Scale (RASS) greater than or equal to a score of -2 or greater.

Exclusion Criteria--

1. Hemodynamically unstable as determined by clinical care team (including but not limited to: oxygen saturation <90%, below target range of mean arterial pressure despite vasoactive or mechanical support, prone positioning, use of mechanical assist device (such as the intra-aortic balloon pump [IABP] or ventricular assist device [VAD]), active management of intracranial hypertension with abnormal intracranial pressure, spinal precautions, uncontrolled seizures, unstable major fracture, large open surgical wound, known controlled active bleeding).
2. Unable to utilize the VitalGo Total Lift BedTM (TLB, Catalog No. V5, Miramar FL) (e.g., height restrictions [>228 cm], weight restrictions [>425 lbs])
3. Pregnant or breast feeding.
4. Anticipated transfer to another hospital within 72 hours.
5. Not anticipated to survive more than 24 hours.
6. Unable to obtain informed consent from either patient or legally authorized representative (LAR).
7. Patients in the ICU but not on ECMO upon enrollment.
8. Patients actively awaiting transplant (heart/lung) without potential for weaning from ECMO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Timing of exercises | From enrollment to 3-month follow-up
  Time spent exercising per each session of rehabilitation program

SECONDARY OUTCOMES:
Mobility | From enrollment to 3-month follow-up
  Maximum Heart Rate (bpm)
Mobility | From enrollment to 3-month follow-up
  Blood Pressure (mmHg)
Mobility | From enrollment to 3-month follow-up
  Respiratory Rate (bpm)
Mobility | From enrollment to 3-month follow-up
  Borg Rating of Perceived Exertion (RPE)--measured on a scale from 6 to 20, where 6 represents "no exertion at all" and 20 represents "maximal exertion"
Mobility | From enrollment to 3-month follow-up
  Steps taken in one minute
Mobility | From enrollment to 3-month follow-up
  Time spent standing away from bed (minutes)
Function | From enrollment to 3-month follow-up
  Functional Independence Measure (FIM) from Activities of Daily Living (ADL). Each ADL will be graded per the FIM Instrument using the disability measure definitions from Total Assistance to Complete Independence.
Resistance Training | From enrollment to 3-month follow-up
  Repetitions will be counted and documented per session per exercise. Grip strength will be tested using a hand dynamometer. The subject will be seated with their elbows at his/her side and flexed at right angles, and their wrists will be at a neutral position. The grip strength of the dominant hand will be tested as the average of three trials

OTHER OUTCOMES:
Quality of Life (QOL) | From enrollment to 3-month follow-up
  The Patient-Reported Outcomes Measurement Information System-29 is a validated and reliable questionnaire that assesses seven health domains: physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. This profile measurement using a standardized T-score system, where scores are interpreted relative to the general US population, with a mean of 50 and a standard deviation of 10; higher scores generally indicate greater impairment in most domains, except for physical function and social participation where higher scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Sousse, PhD, MBA, Principal Investigator — Institute for Extracorporeal Life Support
Locations (1):
- Methodist Healthcare System, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang D, Lim J, Kim BG, Nam H, Kim Y, Kang E, Kim S, Shim S, Lee M, Yoon J, Lee H, Shin SH, Park HY, Cho J. Psychometric validation of the Korean Patient-Reported Outcome Measurement Information System (PROMIS)-29 Profile V2.1 among patients with chronic pulmonary diseases. J Thorac Dis. 2021 Oct;13(10):5752-5764. doi: 10.21037/jtd-21-591. PMID 34795924
- [Background] Fisher CJ, Namas R, Seelman D, Jaafar S, Homer K, Wilhalme H, Young A, Nagaraja V, White ES, Schiopu E, Flaherty K, Khanna D. Reliability, construct validity and responsiveness to change of the PROMIS-29 in systemic sclerosis-associated interstitial lung disease. Clin Exp Rheumatol. 2019 Jul-Aug;37 Suppl 119(4):49-56. Epub 2019 Sep 4. PMID 31498073
- [Background] Eggmann S, Verra ML, Luder G, Takala J, Jakob SM. Effects of early, combined endurance and resistance training in mechanically ventilated, critically ill patients: A randomised controlled trial. PLoS One. 2018 Nov 14;13(11):e0207428. doi: 10.1371/journal.pone.0207428. eCollection 2018. PMID 30427933
- [Background] Hayes K, Holland AE, Pellegrino VA, Young M, Paul E, Hodgson CL. Early rehabilitation during extracorporeal membrane oxygenation has minimal impact on physiological parameters: A pilot randomised controlled trial. Aust Crit Care. 2021 May;34(3):217-225. doi: 10.1016/j.aucc.2020.07.008. Epub 2020 Oct 7. PMID 33039302
- [Background] Hayes K, Holland AE, Pellegrino VA, Mathur S, Hodgson CL. Acute skeletal muscle wasting and relation to physical function in patients requiring extracorporeal membrane oxygenation (ECMO). J Crit Care. 2018 Dec;48:1-8. doi: 10.1016/j.jcrc.2018.08.002. Epub 2018 Aug 7. PMID 30118978
- [Background] Batycka-Stachnik D, Piwoda A, Darocha T, Spiewak M, Kosinski S, Jarosz A, Hymczak H, Sanak T, Galazkowski R, Piatek J, Konstanty-Kalandyk J, Drwila R. Problems and challenges in the early period of rehabilitating patients with severe hypothermia treated using ecmo support. Wiad Lek. 2016;69(3 pt 2):489-494. PMID 27717931
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337